CLINICAL TRIAL: NCT02866240
Title: Safety and Therapeutic Measures of Cathodal Transcranial Direct Current Stimulation (Tdcs) in Patients With Refractory Focal Epilepsy
Brief Title: Safety and Therapeutic Measures of Tdcs in Patients With Refractory Focal Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroelectrics Corporation (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other); Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCHEpilepsy
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single arm (Experimental): Cathodal Transcranial Direct Current Stimulation (tDCS)
  Interventions: Device: Cathodal Transcranial Direct Current Stimulation (tDCS).

INTERVENTIONS:
Device: Cathodal Transcranial Direct Current Stimulation (tDCS). — Transcranial direct current stimulation (tDCS) is a form of neurostimulation which uses constant, low current delivered to the brain area of interest via electrodes on the scalp.

SUMMARY:
This is a single site, non-randomized, prospective, open-label, interventional pilot/feasibility study. Patients recruited will have medically-refractory focal neocortical epilepsy, defined on the basis of presence of focal spikes and (if available) focal seizure onsets originating from the lateral cortical surface of any lobe. All patients and referring physicians will be requested to maintain their current antiepileptic drugs throughout the study with changes after enrollment permitted only to maintain pre-enrollment drug levels, or if clinically necessary. The primary outcome measure will be the change in seizure frequency (seizures/week) as compared to baseline.

Patients with medically-refractory neocortical epilepsy will receive cathodal tDCS administered to the seizure focus for 10 sessions over a 2-week period with the allowance of make-up sessions in week three. Subjects will be evaluated at baseline, during the stimulation sessions, and 8 weeks after the completion of the tDCS visits

DETAILED DESCRIPTION:
Noninvasive neurostimulation techniques include Transcranial magnetic stimulation (TMS) and Cathodal Transcranial Direct Current Stimulation (tDCS). Of these, tDCS is uniquely suited to mass distribution and treatment, even at home, as it is lightweight, portable, inexpensive and has a favorable safety profile. In tDCS, a low intensity (1-2 mA) unidirectional electrical current is applied to the scalp to influence underlying cortical excitability. Some small preliminary studies suggest that cathodal tDCS may suppress epileptic seizures. However, a well-powered randomized-controlled trial demonstrating convincing proof of efficacy has not been conducted. This study is intended to test whether tDCS reduces seizures in patients with intractable focal neocortical epilepsy. The hypothesis is that repeated daily sessions of cathodal tDCS will lead to a clinically significant decrease in seizures in this population. Successful completion of this pilot study will be an essential first step toward a larger placebo-controlled trial with the goal of establishing cathodal tDCS as a novel, non-invasive and inexpensive treatment for drug-resistant seizures, and will provide the critical data needed for an application to obtain FDA approval for the use of tDCS in the treatment of drug-resistant epilepsy.

tDCS is a painless method for focal brain stimulation. tDCS is based on decades-old observations that neuronal firing is modulated by low amplitude electrical direct current (DC). Specifically, when applied to the cerebral cortex, cathodal DC inhibits neuronal firing. The mechanisms by which cathodal DC reduces neuronal firing likely relate to hyper-polarization of the soma membrane which occurs when the apical dendrites neuron are oriented toward the cathode in a constant electric field. The practical application of tDCS is simple: low amplitude DC is administered via scalp electrodes such that the cerebral cortex is exposed to cathodal DC beneath one of the electrodes, and the return (anodal) electrodes can be placed anywhere else on the body, or in more complex arrangements to minimize currents at any one site. tDCS methods have also recently been adapted to rats for work with disease models showing success with seizure suppression. Numerous of tDCS studies have demonstrated the technique to be well tolerated and safe. Direct electrical current stimulation is presently FDA-approved for extracranial use, and FDA applications for tDCS for management of mood disorder and chronic pain are in progress.

tDCS units are also inexpensive and light-weight. The electrical supply can be derived from conventional 9-volt batteries. The scalp electrodes can be fastened in seconds. tDCS can be combined easily with other therapies, such as those that may be required for resuscitation of an acutely-injured patient. tDCS is presently under investigation as a treatment for epilepsy, where excess cortical excitability is a prominent feature of the disease process, and where neuronal inhibition may be beneficial. Thus for epilepsy, tDCS may offer a practical non-pharmacologic therapy for the large minority, approximately 35%, of patients whose seizure cannot be controlled by medication.

The tDCS stimulator used in this clinical study is the STARSTIM device (Neuroelectrics, Inc). STARSTIM is capable of recording EEG before, during and after tDCS stimulation, and will not only allow for a detailed understanding of the tDCS-induced effect on neural activity, but may eventually serve as a guidance to fine-tune the stimulation parameters and improve the tDCS protocol based on the developmental, behavioral, dynamical, and disease state through closed-loop systems.

Starstim device is remotely controlled using NIC software that stands for Neuroelectrics Instrument Controller (NIC). This application will allow physicians to configure the study protocol with all the defined parameters. The provided version of software will only enable to apply tDCS protocols to the subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* 9 years old or older
* An established diagnosis of medically-refractory neocortical epilepsy (as determined by the referring clinician), with a clearly defined seizure focus.
* Diagnosis of epilepsy with focal seizures with or without secondary generalization (International League Against Epilepsy classification). Diagnosis established by clinical history and an electroencephalogram consistent with localization-related epilepsy.
* Continued seizures despite adequate dosage in trials of at least 2 or more antiepileptic medications within approximately the last 3 years.
* At least one clearly identified and localizable epileptogenic zone from which 80% or more seizures arise, as defined by the referring clinician.
* Currently on 1-4 anti-epileptic drugs (AEDs) with no changes in antiepileptic drug doses in the 3 weeks prior to enrollment in the study and no planned dose changes during the trial and through the primary endpoint
* A clinical or research MRI scan that is suitable for navigated brain stimulation (NBS) and generation of electrical fields
* A reported average of at least 3 seizures per month (focal or secondarily generalized) over the three months prior to enrollment, and a minimum of 4 seizures recorded during the 8-week baseline period, with no 21-day seizure-free period during the 8 week baseline
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study. All female participants of child bearing age are required to have a pregnancy test. Additionally, all females of childbearing potential will be required to use an effective method of birth control including: oral hormonal contraceptives; implanted hormonal contraceptives, diaphragm with spermicide; condoms; intra-uterine device; abstinence.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Uncertainty regarding the diagnosis of medically-refractory epilepsy.
* History of Non-epileptic or psychogenic seizures, Primary generalized seizures, Status epilepticus in the last 12 months, Suspicion for or a significant history of syncope, Coexisting significant medical condition that is not in good control, Progressive neurologic disease, Progressive brain disorders, Serious systemic diseases, Symptomatic cerebrovascular disease, Cardiac disease, Chronic skin disease or Damaged skin on scalp that would interfere with tDCS stimulation.
* Any cranial metal implants (excluding dental fillings) or medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagus nerve stimulator).
* Previous surgeries opening the skull.
* Active or recent substance abuse or dependence within the past year.
* No medication is an absolute exclusion from tDCS/TMS. Medications will be reviewed and a decision about inclusion will be made based on the following: patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other central nervous system (CNS) active drugs. The published TMS guidelines review of medications to be considered with TMS will be taken into consideration.
* Any condition that makes the subject, in the opinion of the investigator, unsuitable for the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Seizure frequency in patients with intractable focal neocortical epilepsy using cathodal tDCS. | 8 weeks
  Seizure frequency relative to pre-treatment baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children´S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided